CLINICAL TRIAL: NCT02941068
Title: Prophylactic Annti-fungal Treatment in Severe Sepsis Patients With Perforations in SICU
Brief Title: the Influence of Prophylactic and Empirical Anti-fungal Treatment in Severe Sepsis Patients With Perforations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Principal Investigator, Gao Tao, Clinical Professor, Nanjing PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012NLY032
Record Dates: First submitted 2016-10-15; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Intra-abdominal Perforation
Keywords: severe sepsis; intra-abdominal perforation; surgical intensive care unit; fungal infection; prophylactic anti-fungal treatment
MeSH Terms: conditions — Sepsis; Mycoses | interventions — Fluconazole; Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylactic group (Experimental): Patients would received intravenous fluconazole (loading dose 800 mg, then 400 mg/day) or caspofungin (loading dose 70 mg, then 50 mg/day) if patients had organ failure or renal or liver dysfunction during the immediately surgery. The antifungal treatment would continue for 5 to 7 days.
  Interventions: Drug: fluconazole and caspofungin
- Empirical group (No Intervention)

INTERVENTIONS:
Drug: fluconazole and caspofungin
  Arms: Prophylactic group

SUMMARY:
This prospective intended to observe the influence of prophylactic and empirical anti-fungal treatment on Severe Sepsis patients with perforations. With the consent of patients' legal guardian for prophylactic use of antifungal agents, patients were divided into two groups: prophylactic group and Empirical group.

DETAILED DESCRIPTION:
Intra-abdominal perforation is the high risk of fungal infection. The flora in digestive tract would colonize and go to the blood to develop severe bacteria and fungal infection in intra-abdominal perforation and about one-third of patients with gastrointestinal perforations or anastomotic leakages in ICU develop intra-abdominal fungal infection. In particular, the severe sepsis arisen from these infections could further increase the mortality. However, empiric/preemptive treatment in most studies failed to improve the prognosis and few of the studies that addressed the influence of prophylactic anti-fungal treatment in patients with GI Perforation.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥16 years
2. the time between gastrointestinal perforations or anastopmotic leakage(s) after abdominal surgery and entering ICU within 6 hours
3. ICU stay of at least 5 days
4. APACHE Ⅱ score within 24 hours of randomization of 16 or more
5. severe sepsis
6. written informed consent -

Exclusion Criteria:

1. documented fungus before gastrointestinal perforations/anastopmotic leakage(s) ongoing antifungal treatment before the study;
2. fluconazole/caspofungin allergy;
3. pregnant of lactating woman;
4. life expectancy of 48 hours or less. -

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2012-03; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
all cause mortality | six months

SECONDARY OUTCOMES:
fungal infection | six months
  An blood specimen and abdominal drainage fluids if available were obtained for microbiological culture at the time of the gastrointestinal perforations and intra-abdominal specimen was collected at the time of the immediately surgery. All specimens were also obtained 1st, 3rd, 5th, 7th day after perforations and thereafter at 3 days intervals.

CONTACTS AND LOCATIONS:
Overall Officials: gao tao, ph.d, Principal Investigator — Nanjing PLA General Hospital; cao chun, ph.d, Study Director — Nanjing PLA General Hospital; shi jialiang, ph.d, Principal Investigator — Nanjing PLA General Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Montravers P, Dupont H, Gauzit R, Veber B, Auboyer C, Blin P, Hennequin C, Martin C. Candida as a risk factor for mortality in peritonitis. Crit Care Med. 2006 Mar;34(3):646-52. doi: 10.1097/01.CCM.0000201889.39443.D2. PMID 16505648
- [Result] Senn L, Eggimann P, Ksontini R, Pascual A, Demartines N, Bille J, Calandra T, Marchetti O. Caspofungin for prevention of intra-abdominal candidiasis in high-risk surgical patients. Intensive Care Med. 2009 May;35(5):903-8. doi: 10.1007/s00134-009-1405-8. Epub 2009 Jan 27. PMID 19172247